CLINICAL TRIAL: NCT02158429
Title: Comparison Study of Three-Dimensional vs. Two-Dimensional Ultrasound in Measures of Maternal and Paternal Bonding
Brief Title: Study of Ultrasound To Increase Parental Bonding in Women With Substance Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hawaii (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Tricia E. Wright, M.D., Assistant Professor, University of Hawaii
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USParentalbonding; 5U54RR014607 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-06-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Substance Use Disorders; Pregnancy
Keywords: substance use disorders; pregnancy; maternal attachment; paternal attachment; three dimensional ultrasound
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 Dimensional ultrasound (Active Comparator): an additional 5-10 minutes of ultrasound using three dimensional technique
  Interventions: Other: 2 dimensional vs. 3 dimensional ultrasound
- 2 dimensional (Active Comparator): an additional 5-10 minutes of ultrasound using standard two-dimensional technique
  Interventions: Other: 2 dimensional vs. 3 dimensional ultrasound

INTERVENTIONS:
Other: 2 dimensional vs. 3 dimensional ultrasound — At the end of a regularly scheduled ultrasound measuring fetal growth an additional 5-10 minute ultrasound will be performed, either in 2-dimensional or 3-dimensional mode

SUMMARY:
1. A randomized trial of 3-dimensional vs. 2-dimensional ultrasound, comparing scores on the Maternal Antenatal Attachment Scale (MAAS), a validated instrument measuring maternal attachment as a marker of maternal bonding. The hypothesis is that 3-dimensional ultrasound is better at eliciting maternal attachment than 2-D
2. To assess changes in maternal confidence to stop using drugs and quit/reduce smoking with 3-D vs. 2-D ultrasound. Again, the hypothesis is that 3-D ultrasound will improve the woman's confidence to stop using substances.
3. To evaluate if 3-D ultrasound improves paternal attachment as measured by pre- and post- scores on the Paternal Antenatal Attachment Scale (PAAS). The hypothesis is that 3-D ultrasound will have a greater effect on PAAS scores than 2-D.

DETAILED DESCRIPTION:
To evaluate whether 3-dimensional ultrasound improves measures of maternal attachment compared with 2-D. As substance-using pregnant women are at high risk for intrauterine growth restriction (IUGR), monthly ultrasounds are indicated (Bhuvaneswar, 2008 and Mattioli, 2010). The women will receive a short questionnaire immediately before and 2 weeks after the examination at 22-32 weeks. We will randomize the women to receive either 2-D or 3-D ultrasound with a cross-over at the next ultrasound (mainly to ensure compliance with the study, as women perceive the 3-D ultrasound to be more desirable). The majority of the survey will be the Maternal Antenatal Attachment Scale (MAAS)(Condon 1993) evaluating feelings towards the fetus, pregnancy, and relationship. In addition, three questions will be added to the questionnaire, as addressed in aim 2, which specifically address confidence in the women's ability to stop using drugs and quit or decrease smoking. The main outcome measure will be comparing the pre/post-ultrasound change in the MAAS in the 3-D vs. 2-D ultrasound groups.

Secondary outcomes such as compliance with prenatal care (missed or rescheduled visits), and substance use (including smoking) are routinely collected on our women at each visit. Additionally, historical controls can be gathered from Path clinic data (previously considered exempt by University of Hawaii Committee on Human Studies on 2/24/10).

Ultrasound exams will be provided by the PI or trained ultrasonographer, using a Phillips HD11 WHC 3 and 4 dimensional ultrasound will be used. The PI is a board certified Obstetrician and Gynecologist and has had special training in the use of 3 and 4 dimensional ultrasound. This exam will be a standardized additional 5-10 minutes added onto the end of the routine scan for growth, to obtain a suitable 2-D or 3-D picture of the face and/or hand. These additional views are routinely done in the community. A 5-minute consultation will be done by the PI after each scan, with an opportunity to ask questions. If a previously undiagnosed fetal anomaly is suspected based on this scan (which is extremely unlikely given that they patient has been previously screened by perinatologists), referral for further perinatology consultation will be made. In the extremely unlikely case this happens, the ultrasounds will be covered by the patient's insurance.

The patients will be followed through their pregnancies to measure compliance with prenatal care. Data collection for the purposes of this study will end with the birth of the child.

If the father of the baby is involved, he would be asked to participate. If he consents to participate, he would complete the paternal equivalent to the MAAS (the PAAS) prior to the ultrasound and two weeks after the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a history of substance use during pregnancy obtaining prenatal care between 24-32 weeks of pregnancy

Exclusion Criteria:

* Women less than 18, incarcerated women, women with fetal anomalies previously diagnosed.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Maternal attachment scores | Immediately following scoring
  Comparing the scores pre-and post ultrasound on the MAAS (maternal antenatal attachment scale) survey.

SECONDARY OUTCOMES:
Self-efficacy scales, self perceived efficacy in quitting substances during pregnancy | immediately
  a self-scored scale pre- and post-ultrasound
Birth Outcomes | At delivery, up to 5 months after enrollment
  Comparing birth outcomes including birth weight, gestational age, substance use, NICU stays between the two groups

OTHER OUTCOMES:
Compliance with prenatal care | Upon birth of child. Up to five months after enrollment
  comparing number of prenatal visits between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Tricia E Wright, MD MS, Principal Investigator — University of Hawaii
Locations (1):
- Path Clinic, Honolulu, Hawaii, United States